CLINICAL TRIAL: NCT00339937
Title: Studies of Human Herpesvirus 8 and Kaposi's Sarcoma in Sicily
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998035; OH98-C-N035
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2020-05

CONDITIONS: Kaposi s Sarcoma (KS)
Keywords: Human Herpes virus 8 (HHV8); Kaposi sarcoma (KS)
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Cases: Adults in Italy with Kaposi's sarcoma
- Controls: Adults in Italy without Kaposi's sarcoma

SUMMARY:
A series of studies will be conducted in Sicily by a collaborative team from the U.S. National Cancer Institute and the University of Palermo to better understand the prevalence and risk factors for the newly discovered human herpes virus 8 (HHV8) and Kaposi s sarcoma (KS), which may be a consequence of HHV8 infection. There are four short-term projects:

1. To determine HHV8 seroprevalence in extant, unlinked sera from informative groups, including homosexual men, persons with sexually transmitted diseases, and in general population groups, particularly the elderly. In addition, HHV8 prevalence and other serological studies may be determined among other adults, particularly those who may be recruited for future studies and those likely to enhance understanding of HHV8 serology.
2. To identify a pediatric syndrome that might be associated with HHV8 infection, HHV8 seroprevalence will be determined in sera from hospitalized children with a wide range of clinical conditions.
3. To determine HHV8 seroprevalence in various regions of Italy and by HLA Class II groups that have been linked to increased (HLA-DR5) or decreased (HLA-DR3) risk of KS, using extant, unlinked sera and data from volunteer bone marrow donors.
4. To conduct a case control study that will identify risk factors for KS among persons who are infected with HHV8 and who manifest anti-HHV8 latent antibodies.

The results of these projects will be summarized for publication in the medical and scientific literature and for the design and prioritization of related projects in the future.

DETAILED DESCRIPTION:
A series of studies will be conducted in Sicily by a collaborative team from the U.S. National Cancer Institute and the University of Palermo to better understand the prevalence and risk factors for the newly discovered human herpes virus 8 (HHV8) and Kaposi s sarcoma (KS), which may be a consequence of HHV8 infection. There are four short-term projects:

1. To determine HHV8 seroprevalence in extant, unlinked sera from informative groups, including homosexual men, persons with sexually transmitted diseases, and in general population groups, particularly the elderly. In addition, HHV8 prevalence and other serological studies may be determined among other adults, particularly those who may be recruited for future studies and those likely to enhance understanding of HHV8 serology.
2. To identify a pediatric syndrome that might be associated with HHV8 infection, HHV8 seroprevalence will be determined in sera from hospitalized children with a wide range of clinical conditions.
3. To determine HHV8 seroprevalence in various regions of Italy and by HLA Class II groups that have been linked to increased (HLA-DR5) or decreased (HLA-DR3) risk of KS, using extant, unlinked sera and data from volunteer bone marrow donors.
4. To conduct a case control study that will identify risk factors for KS among persons who are infected with HHV8 and who manifest anti-HHV8 latent antibodies.

The results of these projects will be summarized for publication in the medical and scientific literature and for the design and prioritization of related projects in the future.

ELIGIBILITY:
Pool of HHV8 seropositive controls.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population based samples of adults from Italy (Southern Italy).
Sampling Method: Probability Sample
Enrollment: 4622 (Actual)
Dates: Start 1998-07-30 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Kaposi Sarcoma (KS) | 5 years
  Kaposi Sarcoma (KS)

CONTACTS AND LOCATIONS:
Overall Officials: Sam M Mbulaiteye, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Universita Degli Studi Di Palermo, Palermo, Italy

REFERENCES:
- [Background] Goedert JJ, Biggar RJ, Melbye M, Mann DL, Wilson S, Gail MH, Grossman RJ, DiGioia RA, Sanchez WC, Weiss SH, et al. Effect of T4 count and cofactors on the incidence of AIDS in homosexual men infected with human immunodeficiency virus. JAMA. 1987 Jan 16;257(3):331-4. PMID 3491911
- [Background] Cottoni F, De Marco R, Montesu MA. Classical Kaposi's sarcoma in north-east Sardinia: an overview from 1977 to 1991. Br J Cancer. 1996 May;73(9):1132-3. doi: 10.1038/bjc.1996.217. PMID 8624276
- [Background] Biggar RJ, Nasca PC, Burnett WS. AIDS-related Kaposi's sarcoma in New York City in 1977. N Engl J Med. 1988 Jan 28;318(4):252. No abstract available. PMID 3336414